CLINICAL TRIAL: NCT06747195
Title: The Impact of Intradermal Methylene Blue Injection on the Quality of Recovery in Patients Undergoing Hemorrhoidectomy: a Multicenter Prospective Cohort Study
Brief Title: The Impact of Methylene Blue on the Quality of Recovery in Patients Undergoing Hemorrhoidectomy
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Weifang People's Hospital (Other); Heze Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: Kyll-202405（ZX）-041-3
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Hemorrhoidectomy; Postoperative Analgesia
Keywords: Hemorrhoidectomy; Methylene blue; Quality of recovery; Analgesia; Prospective Cohort Study
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the MB Group: a subcutaneous injection of 0.1% MB (1% MB 2 ml + 1% ropivacaine 5 ml + 0.9% saline 13 ml) will be administered with a skin test needle at the edge of the perianal incision
- the ketorolac group: Patients in the ketorolac group will receive 30 mg of intravenous ketorolac ( Shandong New Times Pharmaceutical Co., Ltd, 1ml:30mg) at the beginning of the procedure.

SUMMARY:
Classical hemorrhoidectomy is known to be linked with significant postoperative pain, which can result in patient discomfort, extended hospital stays, and increased costs. The Quality of Recovery (QOR) score serves as an objective measure of patient-centered general health status following surgery and anesthesia. The latest version, QOR-15, is known for its time-efficiency, high rate of response, and completion, and has been validated in patients undergoing a range of surgical procedures.

Methylene blue (MB) is a water-soluble thiazine dye used to treat various conditions and has been found to have a unique analgesic property through the temporary disruption of anal sensory nerve terminals in patients. Studies conducted in Singapore and China have shown that perianal intradermal injection of MB provides temporary pain relief after hemorrhoidectomy and lateral anal sphincterotomy. However, there is limited published information regarding the impact of MB on the quality of recovery in anorectal surgery. This study aims to evaluate the effect of intradermal MB combined with ropivacaine injection on the quality of recovery for patients undergoing hemorrhoidectomy.

Study population Patients with symptomatic third- and fourth-degree hemorrhoids who are undergoing hemorrhoidectomy under spinal anesthesia and are admitted to the hospitals (145 for each group) will be prospectively enrolled in this study. Before participating, all patients or their caregivers will provide written informed consent. The protocol for this study has been approved by the Ethical Committee of Qilu Hospital of Shandong University with the protocol number Kyll-202405-041-2.

Intervention A standardized spinal anesthesia technique will be utilized, and between 7-9 mg of ropivacaine (Shijiazhuang Siyao Co., Ltd, 10ml:100mg) will be intrathecally injected between the L3 through L5 intervertebral spaces. All patients will undergo hemorrhoidectomy by colorectal surgeons with senior professional titles according to standard techniques. The postoperative analgesia regimen, with or without MB (Jichuan Pharmaceutical Group Co., LTD., 2ml: 20mg), will be determined at the discretion of the colorectal surgeon.

Data collection Clinical data, including age, sex, acute complications and total hospitalization cost, will be collected from the enrolled patients. The QOR-15 score will be calculated for all patients. Over a 6-month follow-up period, complications and the Wexner score for postoperative fecal incontinence will be recorded through telephone interviews.

Outcome measures The primary goal of this study is to evaluate the quality of recovery using the QOR-15 questionnaire, a comprehensive measure of recovery after surgery that assesses five dimensions: physical comfort (5 items), physical independence (2 items), emotional state (4 items), psychological support (2 items), and pain (2 items). Each item is rated on an 11-point scale based on its frequency on the questionnaire (higher scores indicate greater frequency for positive items and less frequency for negative items). The total score ranges from 0 (poorest recovery quality) to 150 (best recovery quality). Patients will complete the QOR-15 questionnaire at three time points: the day before surgery, postoperative day 1, and postoperative day 2 (between 4 pm and 6 pm). The postoperative day 1 score is the primary outcome of interest.

Additional assessments included the following:

The study will collect data on the Visual Analogue Score of pain at multiple time points (postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 7, postoperative day 14), total hospitalization costs, dosage of analgesics three days and fourteen days after surgery, pain leading to unscheduled hospital returns or stay, and various complications such as urinary retention, fecal incontinence, itch and perianal paresthesia, secondary bleeding, perianal infection, poor wound healing at different postoperative time points (postoperative day 1, postoperative day, 1 month postoperative, 3 months postoperative, 6 months postoperative). Additionally, the Wexner score for postoperative fecal incontinence will be recorded at 1 month and 3 months postoperative.

DETAILED DESCRIPTION:
Classical hemorrhoidectomy is often associated with significant postoperative pain, leading to patient discomfort, prolonged hospital stays, and increased costs. The Quality of Recovery (QOR) score serves as an objective measure of patient-centered general health status following surgery and anesthesia. The QOR score allows for the evaluation of various aspects of a patient's recovery experience, including pain, physical comfort, emotional well-being, and the ability to perform daily activities. The latest version, QOR-15, is known for its time-efficiency and high completion rate, making it a valuable tool for assessing patient recovery after surgery and anesthesia.

. Moreover, the QOR-15 has been validated in patients undergoing a wide range of surgical procedures, making it a versatile and reliable measure of postoperative recovery across different medical contexts.

Methylene blue (MB) is a water-soluble thiazine dye that has been utilized to treat various medical conditions. It has been found to possess unique analgesic properties through the temporary disruption of anal sensory nerve terminals in patients. Research conducted in Singapore and China has shown that perianal intradermal injection of MB can offer temporary pain relief following procedures such as hemorrhoidectomy and lateral anal sphincterotomy. This suggests that MB may have potential applications in managing postoperative pain in certain surgical settings. Furthermore, additional studies have demonstrated that individuals suffering from severe anal pruritus (intractable anal pruritus) exhibited improved symptom scores following intradermal injection of methylene blue (MB). This suggests that MB may offer therapeutic benefits for individuals experiencing challenging symptoms of anal pruritus.

The use of methylene blue (MB) for post-hemorrhoidectomy analgesia is still a topic of debate due to certain drawbacks. For instance, there is a latency period of 4-6 hours for MB to exert its analgesic effect after subcutaneous injection, during which the patient may experience burning pain as MB destroys the nerve myelin sheath. Moreover, the use of MB in high concentrations may lead to adverse effects such as anal sensation incontinence and perianal necrosis. Given these potential risks, the study aims to evaluate the effect of intradermal MB combined with ropivacaine injection on Quality of Recovery (QOR) for hemorrhoidectomy patients. The primary hypothesis is that the QOR-15 on postoperative day 1 in patients receiving intradermal MB combined with ropivacaine injection for analgesia will be superior to that in patients receiving intravenous ketorolac for analgesia. This study aims to provide valuable insights into the efficacy and safety of this combined approach for post-hemorrhoidectomy analgesia.

Intervention In the study, a standardized spinal anesthesia technique will be used, and intrathecal injection of between 7-9 mg of ropivacaine (Shijiazhuang Siyao Co., Ltd, 10ml:100mg) will be administered between the L3 through L5 intervertebral spaces. All patients will undergo hemorrhoidectomy by colorectal surgeons with senior professional titles, following standard techniques. The postoperative analgesia regimen, with or without MB ( Jichuan Pharmaceutical Group Co., LTD., 2ml: 20mg), will be at the discretion of the colorectal surgeon. For patients receiving MB, a subcutaneous injection of 0.1% MB (1% MB 2 ml + 1% ropivacaine 5 ml + 0.9% saline 13 ml) will be administered with a skin test needle at the edge of the perianal incision in the MB Group. Patients in the ketorolac group will receive 30 mg of intravenous ketorolac ( Shandong New Times Pharmaceutical Co., Ltd, 1ml:30mg) at the beginning of the procedure. Additional intravenous doses of 30 mg ketorolac may be administered for in-patients, or discharged patients may receive a 10 mg ketorolac pill (Shandong New Times Pharmaceutical Co., Ltd, 10mg) orally if they experience moderate to severe postoperative pain (with a VAS score greater than 3). It is important to note that the maximum daily dose of ketorolac should not exceed 120 mg for intravenous use and 40 mg for oral use. This approach allows for the assessment of the efficacy of intravenous ketorolac for postoperative analgesia in comparison to the intradermal MB combined with ropivacaine injection.

Data collection The study will collect clinical data from enrolled patients, including age, sex, and acute complications such as urinary retention and secondary bleeding. Additionally, the duration of postoperative hospital stay, total hospitalization cost, and the QOR-15 score will be calculated for all patients. During a 6-month follow-up period, complications such as fecal incontinence, itch and perianal paresthesia, perianal infection, and poor wound healing will be recorded through telephone interviews. The Wexner score for postoperative fecal incontinence will also be documented. To ensure data accuracy, extensive training on the study protocol will be provided to all local principal investigators and study staff. Each case will be assigned a researcher who will verify the data against the original medical records to ensure completeness and accuracy. This rigorous approach aims to gather comprehensive and reliable data for the study.

Sample size Based on previous studies that have defined the minimal clinically important difference (MCID) of the QOR-15 as 8, the current study has established the superiority margin for the difference in means between the groups at 8. Our preliminary data indicates that the standard deviation of QOR-15 was 11.2 in the ketorolac group and 8.6 in the MB group. The difference in the mean QOR-15 score between the two groups was 11.1. Based on these findings, the sample size calculation for the superiority test has shown that 260 patients (130 in each group) will be sufficient to demonstrate superiority with a margin of 8, a one-sided significance level of 2.5%, and a power (1-β) of 80%. However, to account for a potential 10% dropout rate, the study will aim to enroll 145 participants in each group.

Statistic The study will analyze categorical variables using Fisher's exact test. For continuous variables, comparisons will be made using independent sample t-tests or Mann-Whitney U tests, depending on the appropriateness of the test for the data distribution. A two-sided p-value of less than 0.05 will be considered statistically significant. Comparisons of QOR-15, VAS, and Wexner scores between different time points will be performed using one-way repeated measures ANOVA. All analysis will be conducted using R software version 3.6.3, Free Statistics software version 1.9, and SPSS version 26. Statistical significance will be set at P < 0.05.

Outcome measures The main goal of this study is to assess the quality of recovery (QOR) using the QOR-15 questionnaire, which is a comprehensive measure of recovery after surgery. The QOR-15 evaluates five dimensions of recovery: physical comfort, physical independence, emotional state, psychological support, and pain. Each dimension consists of a different number of items, and each item is rated on an 11-point scale based on the frequency of the experience reported. A higher score indicates a higher frequency for positive items and a lower frequency for negative items. The total score ranges from 0 (indicating the poorest recovery quality) to 150 (indicating the best recovery quality).

In this study, patients completed the QOR-15 questionnaire at three different time points: the day before surgery, postoperative day 1, and postoperative day 2 between 4 pm and 6 pm. The QOR-15 score on postoperative day 1 is the primary outcome of interest, with the aim of evaluating the quality of recovery on the first day after surgery.

Additional assessments included the following:

This study will assess several outcome measures related to the postoperative period. These measures include: Visual Analogue Scale (VAS) of pain at multiple time points (postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 7, and postoperative day14), duration of postoperative hospital stay, total hospitalization costs, dosage of analgesics three days after surgery and fourteen days after surgery, pain leading to unscheduled hospital returns or stay, various complications at different time points (e.g., urinary retention, fecal incontinence, itch and perianal paresthesia, secondary bleeding, perianal infection, poor wound healing), these are specific postoperative complications that will be monitored at different time points (postoperative day 1, postoperative day 7, 1 month postoperative, 3 months postoperative, and 6 months postoperative). Wexner score for postoperative fecal incontinence at 1 month and 3 months postoperative. These outcome measures will provide a comprehensive evaluation of the postoperative recovery and potential complications following the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mixed hemorrhoids, grade III/ IV hemorrhoids (Goligher's classification), and underwent hemorrhoidectomy under spinal anesthesia; and
* Aged between 18 and 65 years; and
* ASA I or II.

Exclusion Criteria:

* Patients who experienced any ill-effects from previous use of MB or other medications in the protocol (ketorolac, ropivacaine); or
* Patients with diabetes; or
* Alcohol or other addictive drug dependence; or
* Illiteracy, combined with mental system or severe mental illness that prevented completion of the assessment; or
* Patients who are pregnant or breast-feeding; or
* Aspirin and analgesic drugs taken within 2 weeks before surgery; or
* Patients taking selective serotonin reuptake inhibitors (SSRIs); or
* Concurrent additional anorectal diseases (e.g., perianal abscess, anal fistula, fissures, anal incontinence); or
* Patients who are participating in other clinical trials and have not reached the endpoint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This research is a multi-center prospective cohort study conducted at Qilu Hospital of Shandong University, Weifang People's Hospital, and Heze hospital of traditional chinese medicine. All of the patients in the study were of Chinese origin.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Quality of Recovery-15 score on postoperative day 1 | postoperative day 1
  The Quality of Recovery-15 questionnaire, which is a comprehensive measure of recovery after surgery. The QOR-15 evaluates five dimensions of recovery: physical comfort, physical independence, emotional state, psychological support, and pain. Each dimension consists of a different number of items, and each item is rated on an 11-point scale based on the frequency of the experience reported. A higher score indicates a higher frequency for positive items and a lower frequency for negative items. The total score ranges from 0 (indicating the poorest recovery quality) to 150 (indicating the best recovery quality).

SECONDARY OUTCOMES:
the Quality of Recovery-15 on postoperative day 2 | postoperative day 2
The weighted area under the curve (AUC) VAS pain score in the 7 days after surgery | POD1, POD2, POD3, and POD7
postoperative complications | POD1, POD7, 1 month postoperatively, 2 months postoperatively, 3 months postoperatively, 6 months postoperatively
  Various complications at different time points (e.g., urinary retention, fecal incontinence, itch and perianal paresthesia, secondary bleeding, perianal infection, poor wound healing)
Total hospitalization costs | At the time of discharge (assessed up to 5 days)

OTHER OUTCOMES:
The Quality of Recovery-15 score on the day before surgery | the day before surgery
Dosage of analgesics three days after surgery and fourteen days after surgery | within 3 days postoperatively，within 7 days postoperatively
Pain leading to unscheduled hospital returns or stay | up to 1 month postoperatively

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Heze Hospital of Traditional Chinese Medicine, Heze, Shandong
  - Qilu hospital of Shandong University, Jinan, Shandong
  - Weifang People's Hospital, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Yoon S, Joo H, Oh YM, Lee J, Bahk JH, Lee HJ. Validation and clinical utility of the Korean version of the Quality of Recovery-15 with enhanced recovery after surgery: a prospective observational cohort study. Br J Anaesth. 2020 Oct;125(4):614-621. doi: 10.1016/j.bja.2020.06.040. Epub 2020 Jul 21. PMID 32703550
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540